CLINICAL TRIAL: NCT07303231
Title: The Value of Indocyanine Green-guided Near-infrared Fluorescence Technology in Tracing Sentinel Lymph Nodes During Esophagectomy: A Multicenter Prospective Cohort Study
Brief Title: The Value of Indocyanine Green-guided Near-infrared Fluorescence Technology in Tracing Sentinel Lymph Nodes During Esophagectomy
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fujian Medical University Union Hospital (Other)
Collaborators: Henan Cancer Hospital (Other Government); The First Affiliated Hospital of Xiamen University (Other); The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LYNX-ICG
Record Dates: First submitted 2025-01-19; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-05

CONDITIONS: Esophageal Cancer; Sentinel Lymph Node; Lymphadenectomy; Indocyanine Green
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Minimally Invasive Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (ICG group) receiving VATS with near-infrared imaging with indocyanine green to visualize (Experimental)
  Interventions: Drug: Minimally invasive surgery for esophageal cancer using near-infrared indocyanine green fluorescence to visualize the sentinel lymph node
- (Control group) receiving VATS without near-infrared imaging with indocyanine g (No Intervention)

INTERVENTIONS:
Drug: Minimally invasive surgery for esophageal cancer using near-infrared indocyanine green fluorescence to visualize the sentinel lymph node — A multicenter, prospective cohort study will be conducted. Enrolled patients with esophageal squamous cell carcinoma will undergo minimally invasive radical esophagectomy. During surgery, ICG will be injected around the tumor under gastroscopy guidance, and fluorescent lymph nodes will be tracked using a thoracoscopic near-infrared camera. These lymph nodes will be grouped and marked by professional thoracic surgeons, and intraoperative frozen pathology results will be recorded. Subsequent CLND will be performed. The study will collect and analyze patients' clinical information, ICG imaging results, and pathological examination results to explore the effectiveness of the ICG imaging system.
  Arms: (ICG group) receiving VATS with near-infrared imaging with indocyanine green to visualize

SUMMARY:
Sentinel lymph nodes, as the primary site of tumor metastasis, play a pivotal role in assessing patient prognosis and planning subsequent treatment strategies. The investigators plan to conduct a multicenter, prospective cohort study to evaluate the effectiveness of indocyanine green (ICG)-guided near-infrared imaging in tracing sentinel lymph node during esophageal squamous cell carcinoma (ESCC) surgery, compared with the gold standard of complete lymph node dissection (CLND), in detecting metastatic disease. This study aims to address the following core questions:

1. In ESCC patients undergoing surgery, can sentinel lymph node biopsy reduce unnecessary lymph node dissection?
2. In ESCC patients undergoing surgery, can reducing lymph node dissection decrease postoperative complications such as chylothorax and weakened immunity? During the study, ICG will be injected around the tumor under intraoperative gastroscopy guidance, followed by tracking of fluorescent lymph nodes using a thoracoscopic near-infrared camera. Professional thoracic surgeons will group and mark these lymph nodes for intraoperative frozen pathology. Subsequent CLND and routine postoperative pathology will be performed. This study will collect patients' clinical information, ICG imaging results, pathological examination results, and other data for statistical analysis to assess the sensitivity and negative predictive value (NPV) of the ICG imaging system. If the study results support the effectiveness of the ICG imaging system, it has the potential to become an important tool for sentinel lymph node localization and biopsy in future ESCC surgeries, helping to reduce unnecessary lymph node resection and improve surgical efficiency and safety.

Participants will:

1. Undergo minimally invasive ESCC surgery within 2 weeks of enrollment, including the 14th day.
2. Receive ICG injection around the tumor under intraoperative gastroscopy guidance during surgery.
3. Have perioperative, postoperative pathology, and complication information recorded.
4. Undergo standardized follow-up after surgery.

DETAILED DESCRIPTION:
This study will be accepted in esophageal cancer patients with Radical Esophag-ectomy as the research object. The investigators will divide participants into two groups: experimental group for injection of indocyanine green group and control group for injectable in-docyanine green group.The investigators will compare with the accuracy,false positive rate and false negative rate,sensitivity, specificity and related indicators of intraoperative lymph node cleaning,in order to explore the common position of esophageal cancer sentinel lymph node,guidance of esophageal cancer lymph node cleaning thoroughly.

ELIGIBILITY:
Inclusion Criteria:

1. Age and gender: 18-75 years old, male and female unlimited;
2. Preoperative biopsy was pathologically diagnosed as esophageal squamous cell carcinoma;
3. Preoperative combination with neoadjuvant chemoradiotherapy;
4. Surgical resection of esophageal carcinoma under endoscopic selection and intraoperative anastomosis;
5. Heart, lung, liver and kidney functions can tolerate operation;
6. Patients and their family members can understand and are willing to participate in this clinical study and sign the informed consent.

Exclusion Criteria:

1. Allergic to ICG or iodine;
2. Patients with a history of chest surgery or thoracic lymph node dissection;
3. Patients needing emergency surgery;
4. Patients whose tumors involve neighboring organs and need to be removed by combining organs;
5. Patients with tumor recurrence or distant metastasis;
6. Patients who had participated in or were participating in other clinical trials within the previous 4 weeks were included;
7. A history of serious mental illness;
8. Pregnant or lactating women;
9. Patients with other conditions considered by the researcher should not participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy rate of lymph node dissection | 1 week after operation
  According to postoperative pathological results, investigate the detection rate of metastatic lymph nodes using the near-infrared indocyanine green fluorescence imaging system in lymph node dissection for esophageal squamous cell carcinoma

SECONDARY OUTCOMES:
Sensitivity and specificity of lymph node dissection | 1 week after operation
  Sensitivity and specificity of lymph node dissection of each arm（according to postoperative pathology）
The number of lymph nodes | 1 week after operation
  The number of lymph nodes between the both groups
False positive rate of lymph node dissection | 1 week after operation
  False positive rate of lymph node dissectionof each arm（according to postoperative pathology）
False negative rate of lymph node dissection | 1 week after operation
  False negative rate of lymph node dissection of each arm（according to postoperative pathology）

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No